CLINICAL TRIAL: NCT02625740
Title: Use of Local Ultrasound to Enhance Local Paclitaxel Delivery Effect After Femoro-popliteal Percutaneous Transluminal Angioplasty in Patients With Critical Limb Ischemia: the PACUS Trial
Brief Title: Ultrasound to Enhance Paclitaxel Uptake in Critical Limb Ischemia: the PACUS Trial
Acronym: PACUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Roberto Gandini, Medical Doctor, University of Rome Tor Vergata
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tor Vergata University
Record Dates: First submitted 2015-11-30; First posted 2015-12-09 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Peripheral Arterial Disease, Angioplasty
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study group (Experimental): After crossing the lesion with a guidewire, patients will be treated with intravascular high intensity, low-frequency ultrasound followed by local administration of liquid mixture of Paclitaxel and Iopromide-370 with predetermined dosage of 1.0 µg/mm
  Interventions: Device: Local exposition of target lesion to high intensity, low-frequency ultrasound; Device: Flow occlusion with an angioplasty balloon; Drug: Local Paclitaxel infusion; Procedure: Angiographic control
- Control group (Active Comparator): After crossing the lesion with a guidewire, patients will be treated with drug eluting ballon angioplasty with the In.Pact Admiral ballon (Medtronic)
  Interventions: Device: drug eluting ballon angioplasty; Procedure: Angiographic control

INTERVENTIONS:
Device: Local exposition of target lesion to high intensity, low-frequency ultrasound — Target lesion was exposed to 60 seconds of high intensity, low-frequency ultrasound generated by the Genesis™ system ( CardioProlific Inc., Hayward, CA). The ultrasound catheter is removed after the exposition.
  Arms: Study group
Device: drug eluting ballon angioplasty — Target lesion was treated with an angioplasty, performed using the INPACT Admiral drug eluting ballon (Medtronic)
  Arms: Control group
Device: Flow occlusion with an angioplasty balloon — Inflation of a 2 cm long balloon catheter Admiral (Medtronic) , located distally to the treatment area, in order to obtain a flow cessation
  Arms: Study group
Drug: Local Paclitaxel infusion — Paclitaxel in a mixture with contrast medium at 1.0 µg/mm³ concentration was delivered to the treatment area for 60 seconds. The column of the Paclitaxel mixture filling the vessel was observed under the fluoroscopy and sustained during 60 seconds. The Paclitaxel /contrast medium mixture was then aspired with a 50 cc syringe and the distal balloon was deflated.
  Arms: Study group
Procedure: Angiographic control — A final angiographic control was performed with injection of 10 cc of contrast medium and compared with the pre-procedural one.

SUMMARY:
The PACUS Trial was a single center, single blinded, randomized trial designed to evaluate the safety and efficacy of intravascular percutaneous catheter-delivered ultrasound energy to improve local Paclitaxel delivery effects in critical limb ischemia patients due to femoral-popliteal artery disease.

DETAILED DESCRIPTION:
Study design The PACUS Trial was a single center, single blinded, randomized trial designed to evaluate the safety and efficacy of intravascular percutaneous catheter-delivered high intensity, low-frequency ultrasound utilizing CardioProlific Genesis™ System to improve local paclitaxel delivery effect in patients with CLI due to femoral-popliteal calcific lesions and occlusions. The protocol was approved by a Local Review Boards and the Institutional Ethics Committee. All patients provided written informed consent before enrollment. The trial was conducted in accordance with the declaration of Helsinki.

Randomization Randomization occurred after successful crossing and pre-dilatation of the target lesion with a standard percutaneous angioplasty balloon without sub-intimal approach and/or flow limiting dissections. Patients were enrolled when a successful angiographic control was performed after PTA pre-dilatation. Subjects were randomly assigned by a computer-generated random sequence (2 blocks in a 1:1 ratio). Randomization was done in advance for all patients and without any stratification. The patients and physicians involved in the follow-up control were blinded to the treatment assignments through the completion of all 6 month follow-up evaluation. Operators were not blinded due to differences in treatment protocol. Twenty eight (28) patients were treated with an intravascular percutaneous catheter-delivered high intensity, low-frequency ultrasound and local Paclitaxel delivery with temporarily blood flow occlusion created by distal occlusion balloon (Study Group), and twenty eight (28) patients were treated with drug eluting balloon with conventional method (Control Group).

ELIGIBILITY:
Inclusion Criteria:

* Rutherford category ≥4
* femoral-popliteal lesion ≥10cm
* successful intraluminal recanalization without need of a stent to obtain a satisfactory angiographic result
* at least one patent below the knee vessel
* patients older than 18 years

Exclusion Criteria:

* Rutherford category < 4
* pregnancy
* known allergies to study medications and materials
* need of sub-intimal approach to perform the recanalization
* target vessel stent release

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with Freedom from clinically driven target lesion revascularization (TLR) and significant restenosis | 6 months follow up
  Freedom from clinically driven target lesion revascularization (TLR) and significant restenosis as determined by digital subtraction angiography at 6 months follow-up
Number of device and procedure related deaths and major adverse clinical events | 1 months follow-up
  Number of device and procedure related death and major adverse clinical events defined as stroke, myocardial infarction, need of surgical revascularization, distal embolization, recurrence of critical limb ischemia.

SECONDARY OUTCOMES:
Percentage of Intraoperative Technical success | Intraoperative
  Percentage of Technical success (Patients with technical success/Total population) was defined as successful recanalization of the target vessel with ≤30% residual stenosis after the procedure
Number of participants with Clinically driven target lesion revascularization | 12 months follow up
  Number of participants with Target lesion revascularization, defined as any repeat surgical or percutaneous interventions of the target lesion due to loss of patency as evaluated by DSA
Number of participants with clinical improvement | 12 months follow up
  Number of participants with Clinical improvement, defined as freedom from target limb amputation, target vessel revascularization, and increase in Rutherford class.
Number of Death and major adverse clinical events | 12 months follow up
  Number of death and major adverse clinical events included stroke, myocardial infarction, need of surgical revascularization, distal embolization, recurrence of critical limb ischemia.